CLINICAL TRIAL: NCT03416634
Title: Exercise is Medicine (EIM): A Quality Improvement and Pragmatic Trial at Emory Seavey Internal Medicine Clinic
Brief Title: Exercise is Medicine at Emory Seavey Internal Medicine Clinic
Acronym: EIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Sharon Horesh Bergquist, Assistant Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00101370
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Physical Activity
Keywords: Health promotion; Behavioral research; Preventive medicine; Obesity; Cardiovascular disease
MeSH Terms: conditions — Motor Activity; Obesity; Cardiovascular Diseases | interventions — Amyloid; Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: 90 participants will use a wearable device and 90 will use a smartphone app to track activity. These groups will be further randomized to receive an automated motivational intervention, or a personalized motivational intervention or no additional intervention; each study arm will have 30 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- App Alone (Active Comparator): Participants randomized to use the Microsoft Band app to track daily activity
  Interventions: Behavioral: App
- App Plus Automated Motivational Message (Experimental): Participants randomized to use the Microsoft Band app to track daily activity, and to receive automated, motivational text messages
  Interventions: Behavioral: App; Behavioral: Automated Motivational Message
- App Plus Personalized Motivational Message (Experimental): Participants randomized to use the Microsoft Band app to track daily activity, and to receive personalized, motivational text messages
  Interventions: Behavioral: App; Behavioral: Personalized Motivational Message
- Wearable Device Alone (Active Comparator): Participants randomized to use the Garmin vivofit 3 wearable device to track daily activity
  Interventions: Behavioral: Wearable Device
- Wearable Device Plus Automated Motivational Message (Experimental): Participants randomized to use the Garmin vivofit 3 wearable device to track daily activity, and to receive automated, motivational text messages
  Interventions: Behavioral: Wearable Device; Behavioral: Automated Motivational Message
- Wearable Device Plus Personalized Motivational Message (Experimental): Participants randomized to use the Garmin vivofit 3 wearable device to track daily activity, and to receive personalized, motivational text messages
  Interventions: Behavioral: Wearable Device; Behavioral: Personalized Motivational Message

INTERVENTIONS:
Behavioral: App — The Microsoft Band app can be installed for free on compatible smartphones. The app can be used to track steps while the phone is with the participant (such as in a pocket). Participants can synchronize their device with the study app to give permission to share physical activity level with the study team. Daily physical activity will be tracked for 24 weeks.
  Arms: App Alone; App Plus Automated Motivational Message; App Plus Personalized Motivational Message
Behavioral: Wearable Device — A Garmin vivofit 3 fitness device will be provided for free to participants randomized to this study arm. This wearable device tracks daily activity and gives reminders to move after an hour of inactivity. The battery lasts for one year and the device is water resistant. Participants can synchronize their device with the study App to give permission to share physical activity level with the study team. Daily physical activity will be tracked for 24 weeks.
  Arms: Wearable Device Alone; Wearable Device Plus Automated Motivational Message; Wearable Device Plus Personalized Motivational Message
Behavioral: Automated Motivational Message — An automated behavioral intervention will be delivered once weekly via an in-app motivational message, over the 12-week intervention period.
  Arms: App Plus Automated Motivational Message; Wearable Device Plus Automated Motivational Message
Behavioral: Personalized Motivational Message — A behavioral intervention will be delivered once weekly via an in-app motivational message adapted to each patient's personalized PA goal progression based on the previous week data from the smartphone activity app (Microsoft band) or the Garmin wearable device over a 12-week intervention period.
  Arms: App Plus Personalized Motivational Message; Wearable Device Plus Personalized Motivational Message

SUMMARY:
Implementation of physical activity promotion in routine health care delivery is low because of multiple barriers including insufficient health system support, care team coordination, and scarcity of community resources for referring patients and technology tools for sustaining lifestyle changes. This study is a pilot project to test the feasibility of implementing a physical activity promotion protocol, including routine evaluation of patient's physical activity levels and provision of educational material in the clinical workflow. Physically inactive adult patients with at least one documented cardiovascular disease risk factor will be invited to participate in physical activity intervention. Patients will be randomized to receive a wearable device or a smartphone app to objectively monitor their physical activity. Participants will be further randomized to receive automated motivational text messages, or a personalized motivational message, or no messages. Participants will be followed through the 12 week intervention period and an additional 12 weeks with no intervention.

DETAILED DESCRIPTION:
Improving and maintaining health-enhancing levels of physical activity (PA) leads to reductions in the metabolic, hemodynamic, body composition, epi-genetic and functional status risk factors that heavily contribute to the development of many non-communicable chronic diseases. As such, PA has a significant role, in many cases comparable or superior to drug interventions, in the prevention and treatment of more than 40 diseases such as obesity, heart disease, diabetes, hypertension, cancer, depression, anxiety, arthritis, and osteoporosis.

While conceptually simple, implementing clinical-community linkages for PA promotion is hindered by barriers at multiple levels such as inadequate training and self-efficacy among health care providers (HCPs), insufficient health system support and care team coordination, and scarcity of certified community resources for referring patients. The challenge for HCPs and health systems is how to operationalize, standardize, and implement PA promotion in a cost-effective and innovative fashion.

This study is a pilot project to test the feasibility of implementing a physical activity promotion protocol including routine evaluation of patient's physical activity levels and provision of educational material in the clinical workflow of the Seavey Internal Medicine Clinic at Emory University. Physically inactive adult patients with at least one documented cardiovascular disease risk factor (overweight/obesity, dyslipidemia, hypertension, diabetes) but cleared for self-directed exercise by their treating clinician will be invited to participate in physical activity intervention. Patients will be randomized to receive a wearable device (Garmin vivofit 3) or a smartphone app (Microsoft Band) to objectively monitor their physical activity. Participants will be further randomized to receive automated motivational text messages, or a personalized motivational message, or no messages. Participants will be followed through the 12 week intervention period and an additional 12 weeks with no intervention. The researchers will assess changes in objectively-measured physical activity (primary outcome) and explore impact on secondary outcomes including cardiovascular disease (CVD) risk factors (assessed routinely as part of clinical management), as well as self-reported mental health, quality of life and exercise self-efficacy using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* At least one documented cardiovascular disease risk factor
* Not meeting physical activity (PA) guidelines (aerobic and/or muscle-strengthening standards)
* contemplating PA engagement
* Non-wheelchair bound (other assist devices will be acceptable) or major physical limitations for PA
* Cleared for independent PA by their health care provider
* Willingness to participate and provide written informed consent
* Report access to a mobile phone with data plan and/or computer with internet access
* Agrees to not own/use a different PA wearable device during the study period.

Exclusion Criteria:

* Documented unstable angina or myocardial infarction in the past 3 months without having finalized an initial cardiac rehabilitation program;
* Documented end-stage renal disease or life-threatening disease;
* Diagnosed major mental health disorder;
* Alcohol or drug abuse.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity | Baseline through Week 24
  Physical activity will be measured through the Microsoft Band app or with the Garmin vivofit 3. The physical activity of the participants will be monitored during the 12 week intervention period (when some study arms will receive motivational messages) and through 12 additional weeks of follow up.

SECONDARY OUTCOMES:
Change in weight | Baseline through Week 24
  Weight in kilograms will be measured at baseline and throughout the study period.
Change in triglycerides | Baseline through Week 24
  The cardiovascular disease risk factor of dyslipidemia will be assessed by measuring triglycerides at baseline and throughout the study period. Triglycerides above 150 mg/dL are considered high.
Change in total cholesterol | Baseline through Week 24
  The cardiovascular disease risk factor of dyslipidemia will be assessed by measuring total cholesterol at baseline and throughout the study period. Total cholesterol above 200 mg/dL is considered high.
Change in hypertension status | Baseline through Week 24
  The cardiovascular disease risk factor of hypertension will be assessed by measuring blood pressure at baseline and throughout the study period. Blood pressure will be measured as systolic and diastolic millimeters of mercury (mmHg). A blood pressure reading of 140/90 mmHg for a sustained period is considered hypertension.
Change in blood glucose | Baseline through Week 24
  Blood glucose levels will be measured at baseline and throughout the study. Normal fasting blood glucose levels are between 70 and 100 mg/dL.
Change in hemoglobin A1c (HbA1c) | Baseline through Week 24
  HbA1c levels will be measured at baseline and throughout the study. The normal range for HbA1c levels is between 4% and 5.6% of total hemoglobin. Diabetes is diagnosed if HbA1c is greater than 6.5%.
Change in Center for Epidemiologic Studies Depression Scale (CES-D) Score | Baseline, Week 12, Week 24
  Symptoms of depression will be measured with the Center for Epidemiologic Studies Depression Scale (CES-D), National Institute of Mental Health (NIMH). The CES-D asks respondents to indicate how they have felt or behaved in the past week to 20 symptoms of depression, such as "My sleep was restless" and "I was happy". Participants will select from Rarely (<1 day), Some of the time (1-2 days), Occasionally (3-4 days) and Most of the time (5-7 days). Responses are scored from 0 to 3, with reverse scoring for positive items so that 0 corresponds with low symptoms. Total possible scores range from 0 to 60, with higher scores indicating increased symptoms of depression.
Change in Eating Habits Confidence Survey Score | Baseline, Week 12, Week 24
  Self-efficacy to make dietary changes will be measured with the Eating Habits Confidence Survey. This survey asks participants to rate how confident they are that they could motivate themselves to make certain dietary changes for 6 months. The 20-item survey includes statements such as "Eat smaller portions at dinner" and respondents indicate how sure they can do each item on a 5 point scale where 1 = "I know I cannot" and 5 = "I know I can". Total scores range from 20 to 100, where higher scores indicate increased confidence in making dietary changes.
Change in Exercise Confidence Survey Score | Baseline, Week 12, Week 24
  Self-efficacy to make changes in exercise habits will be measured with the Exercise Confidence Survey. This survey asks participants to rate how confident they are that they could motivate themselves to make certain changes to physical activity habits for 6 months. The 12-item survey includes statements such as "Get up early, even on weekends, to exercise" and respondents indicate how sure they can do each item on a 5 point scale where 1 = "I know I cannot" and 5 = "I know I can". Total scores range from 12 to 60, where higher scores indicate increased confidence in making changes to exercise habits.
Change in Social Support and Exercise Survey Score | Baseline, Week 12, Week 24
  The Social Support and Exercise Survey assesses how much support the respondent receives from family members and friends. Participants will rate how often each of the 13 incidents specified occurred in the last three months, rating family and friends separately. Each item is rated on a scale of 1 to 5 where 1 = none and 5 = very often. The responses will be summed to obtain an overall score of the support received from family and friends. Total scores can range from 26 to 130. Scores for particular items are scored in reverse so that higher scores indicate more support.
Change in Short-Form Patient Satisfaction Questionnaire (PSQ-18) Score | Baseline, Week 12, Week 24
  The Short-Form Patient Satisfaction Questionnaire (PSQ-18) asks respondents how much they agree with statements related to the medical care they receive. The 18-item questionnaire includes statements such as "Doctors are good about explaining the reason for medical tests" and "Doctors sometimes ignore what I tell them". Each item is rated from 1 (strongly agree) to 5 (disagree). All items are scored so that high scores reflect satisfaction with medical care. Total scores can range from 18 to 90.
Change in 12-Item Short-Form Health Survey (SF-12) Score | Baseline, Week 12, Week 24
  The 12-Item Short-Form Health Survey (SF-12) asks respondents to rate their health and abilities to do their usual tasks. The SF-12 uses a variety of questions and response options and includes a physical health component summary and a mental health component summary. Scores are reversed, when appropriate, so that a higher value indicates better health. The scale is transformed to have a mean of 50 and a standard deviation of 10; scores above 50 indicate better health than the general US population, while scores below 50 indicate poorer than average health.
Change in 36-Item Short-Form Health Survey (SF-36) Score | Baseline, Week 12, Week 24
  The 36-Item Short-Form Health Survey (SF-36) asks respondents to rate their health and abilities to do their usual tasks. The SF-36 uses a variety of questions and response options and includes 8 subscales (physical functioning, role limitations due to physical health, role limitations due to emotional health, energy/fatigue, emotional well-being, social functioning, pain, and general health). Responses are coded on a scale of 0 to 100 where 0 is the worst possible health and 100 is the most favorable health score. The coded responses will be summed and averaged to obtain a mean score for the entire survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Bergquist, MD, Principal Investigator — Emory University; Roberto Felipe Lobelo, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Paul W. Seavey Internal Medicine Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided